CLINICAL TRIAL: NCT04920747
Title: Interest of the Addition of Docetaxel to Standard Treatment in First-line Advanced HER2 Positive Gastroesophageal Adenocarcinoma in Selective Patients
Acronym: TandHER
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: 2021/622
Record Dates: First submitted 2021-06-04; First posted 2021-06-10 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: HER2-positive Gastric Cancer; Metastatic Cancer; Docetaxel; Trastuzumab
Keywords: docetaxel; trastuzumab; Advanced HER2 Positive Gastroesophageal Adenocarcinoma
MeSH Terms: conditions — Neoplasm Metastasis | interventions — taxane

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- S group: platin-5FU + trastuzumab
- T group: taxanes + platin-5FU + trastuzumab
  Interventions: Drug: Taxane

INTERVENTIONS:
Drug: Taxane — docetaxel or paclitaxel
  Groups: T group

SUMMARY:
The purpose of this retrospective study is to evaluate the efficacy and the safety of trastuzumab + chemotherapies with or without taxanes among HER2-positive advanced gastroesophageal adenocarcinoma patients.

DETAILED DESCRIPTION:
Studies have reported a beneficial role of trastuzumab combined to platin-5-FU based chemotherapy in first-line advanced HER2 positive gastroesophageal adenocarcinoma. However, the effect of taxanes combined with platin-5FU + trastuzumab (TPFT) is understudied.

In this context, the aim of this study is to evaluate the efficacy and the safety of trastuzumab + chemotherapies with or without taxanes among HER2-positive advanced gastroesophageal adenocarcinoma patients.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed non-resectable locally advanced, recurrent, or metastatic adenocarcinoma of the stomach or gastro-esophageal junction;
* tumor samples scored as 3+ on immunohistochemistry or FISH (Fluorescence in situ Hybridization) positive (HER2:CEP17 ratio ≥2);
* measurable disease;
* treated by trastuzumab, platin (cisplatine or oxaliplatine), fluoropyrimidine (5-FU or capecitabine) +/- taxanes (docetaxel or paclitaxel),
* as first-line therapy for advanced gastric cancer.

Exclusion Criteria:

* previous chemotherapy by taxane for metastatic disease,
* previous anti-HER2 therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated between January 2009 and Mars 2021 were included, in 7 centers in Franche-Comte region in France.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Progression free survival | up to 12 years
  PFS will be defined as the time interval between the date of randomization and the date of first progression (local, regional, metastatic, second cancer) or death regardless of the cause. Patients alive without progression will be censored at the time of the latest news

SECONDARY OUTCOMES:
Overall survival | up to 12 years
  OS will be calculated between the date of randomization and the date of death from any cause. . Alive patients or lost to follow-up at the time of the analysis will be censored at the date of last follow-up.
Objective Response Rate | up to 12 years
  Evaluated by RECIST criteria version 1.1
disease control rate | up to 12 years
secondary resectability of primary tumor or metastases in patients with DCR | up to 12 years
Tolerance | up to 12 years
  graded according to National Cancer Institute-Common Terminology Criteria for Adverse Events [NCI-CTCAE] criteria v4.03

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Besancon, Besançon, Franche-Comté, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Orillard E, Henriques J, Vernerey D, Almotlak H, Calcagno F, Fein F, Fratte S, Jary M, Klajer E, Vienot A, Borg C, Kim S. Interest of the Addition of Taxanes to Standard Treatment in First-Line Advanced HER2 Positive Gastroesophageal Adenocarcinoma in Selective Patients. Front Oncol. 2022 Mar 7;12:763926. doi: 10.3389/fonc.2022.763926. eCollection 2022. PMID 35340264